CLINICAL TRIAL: NCT04144738
Title: Clinical Validation of An Optimized Multi-Target Stool DNA (Mt-sDNA 2.0) Test, for Colorectal Cancer Screening "BLUE-C"
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Sample Collection; Stool DNA; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual stool samples will be used to develop and evaluate the performance of biomarker assays to detect cancers and advanced precancerous lesions. Samples may be stored for up to 20 years. These stool samples will be de-identified.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals eligible for CRC Screening: Individuals who are 40 years of age and older, eligible for CRC screening, and scheduled for a screening colonoscopy.
  Interventions: Diagnostic Test: mt-sDNA 2.0 screening test; Diagnostic Test: FIT test; Procedure: Colonoscopy

INTERVENTIONS:
Diagnostic Test: mt-sDNA 2.0 screening test — Stool samples will be collected by the subject for the mt-sDNA screening test.
Diagnostic Test: FIT test — Stool samples will be collected by the subject for the FIT test.
Procedure: Colonoscopy — Subjects will undergo a screening colonoscopy.

SUMMARY:
The primary objective of this study is to assess the sensitivity for colorectal cancer (CRC) and specificity of the mt-sDNA 2.0 test.

DETAILED DESCRIPTION:
Subjects 40 years of age and older scheduled for a screening colonoscopy will be enrolled. Subject will complete the mt-sDNA 2.0 test and the commercially available FIT, followed by completion of a screening colonoscopy. The results of the mt-sDNA screening test and FIT will not be provided to investigators for clinical management of the study subject. Personnel performing the colonoscopy and producing the resulting report and personnel performing histopathologial review of reports or tissue (if applicable) will remain blinded to the results of the mt-sDNA 2.0 screening test results.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for the study:

1. Subject is ≥ 40 years of age at the time of enrollment.
2. Subject presents for a screening colonoscopy per standard of care.
3. Subject has no symptoms or signs that require immediate, or near term, referral for diagnostic or therapeutic colonoscopy.
4. Subject is able and willing to sign informed consent

Exclusion Criteria:

1. Subject has a history of CRC or advanced precancerous lesions.
2. Subject has a diagnosis or medical / family history of any of the following conditions, including:

   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome),
   * Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome"),
   * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis, or Familial Hyperplastic Polyposis.
3. Subject has a diagnosis or personal history of inflammatory bowel disease (IBD) including chronic ulcerative colitis and/or Crohn's disease.
4. Subject has a diagnosis of Cronkhite-Canada Syndrome.
5. Subject has had a positive Cologuard within the previous 2 years, or fecal occult blood test or FIT within the previous 6 months.
6. Subject has undergone a colonoscopy within the previous 9 years with the exception of a failed colonoscopy due to poor bowel preparation. Failed colonoscopy must have been within the past year and without therapeutic intervention.
7. Subject has had overt rectal bleeding within the previous 30 days.
8. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 40 years of age and older who are eligible for CRC screening and scheduled for a screening colonoscopy. 24,000 subjects are targeted to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 26758 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity for CRC with the mt-sDNA 2.0 test | Through study completion, an average of 180 days
Specificity with the mt-sDNA 2.0 test | Through study completion, an average of 180 days

SECONDARY OUTCOMES:
Sensitivity for advanced precancerous lesions | Through study completion, an average of 180 days
Sensitivity for CRC compared to a commercially available fecal immunochemical test (FIT) | Through study completion, an average of 180 days
Sensitivity for advanced precancerous lesions compared to commercially available fecal immunochemical test (FIT). | Through study completion, an average of 180 days
Specificity for no colorectal neoplastic findings | Through study completion, an average of 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, MD, Principal Investigator — Indiana University
Locations (194):
- United States (194):
  - Parkway Medical Center, Birmingham, Alabama
  - Summit Internal Medicine, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - G & L Research, Foley, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - East View Medical Research, LLC, Mobile, Alabama
  - GI Associates of West Alabama, P.C, Tuscaloosa, Alabama
  - Mayo Clinic - AZ, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Southern Arizona VA Health Care System (SAVAHCS), Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, P.A., North Little Rock, Arkansas
  - Fomat Medical Research, Camarillo, California
  - Alliance Research Institute, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Paragon Rx Clinical, Inc., Garden Grove, California
  - United Medical Doctors, Irvine, California
  - Prime Care Clinical Research Center, Laguna Hills, California
  - Gastro Care Institute, Lancaster, California
  - Facey Medical Foundation, Mission Hills, California
  - Knowledge Research Center, Orange, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Palo Alto Veterans Institute for Research, Palo Alto, California
  - SDG Clinical Research, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Paragon Rx Clinical, Inc. - Santa Ana, Santa Ana, California
  - Sansum Clinic, Santa Barbara, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Dream Team Clinical Research, Upland, California
  - New West Physicians, Golden, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Yale University, New Haven, Connecticut
  - Cornerstone Research Institute, Altamonte Springs, Florida
  - Vanguard Clinical Research, Fort Myers, Florida
  - SIMED Health Research, Gainesville, Florida
  - Westside Center of Clinical Research, Jacksonville, Florida
  - Shands Jacksonville Medical Center, Inc - University of Florida Health, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Wr-Msra, Llc, Lake City, Florida
  - Pioneer Clinical Research, Lighthouse PT, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Gastro Health Research, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Imic, Inc., Palmetto Bay, Florida
  - Family Medical Specialists of Florida, PLC, Plant City, Florida
  - Alternative Solutions, LLC, St. Petersburg, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Clinical Trials of Tampa, Tampa, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Augusta University, Augusta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Christie Clinic, LLC, Champaign, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - GI Partners of IL / Avicenna, Downers Grove, Illinois
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Margaret Mary Health, Batesville, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana
  - Deaconess Clinic, Inc., Newburgh, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - PMG Research, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - Digestive Health Center of the Four States, LLC, Galena, Kansas
  - Hutchinson Clinic, Hutchinson, Kansas
  - Ascension Via Christi Hospitals Wichita, Inc, Wichita, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Houma Digestive Health Specialists-CroNOLA, Houma, Louisiana
  - Combined Gastro Research, LLC, Lafayette, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center; Gastrointestinal Associates, Shreveport, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Gastro Health Research, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Harvard, Boston, Massachusetts
  - IQVIA RDS, Inc., Cambridge, Massachusetts
  - Digestive Health Specialists, PC, Chelmsford, Massachusetts
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - University of Massachusetts - Worcester, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Clinical Research Institute of Michigan, LLC, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC (STAR), Jackson, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Methodist Physicians Clinic / CCT Research, Fremont, Nebraska
  - CHI Nebraska, Omaha, Nebraska
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Digestive Health Associates, Reno, Nevada
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Allied Health Clinical Research Organization, LLC, West Long Branch, New Jersey
  - United Health Services Hospitals, Inc., Binghamton, New York
  - VA NY Harbor HCS- Brooklyn Campus, Brooklyn, New York
  - Sing Chan, MD, Flushing, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - Digestive Health Partners, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Department of Family Medicine Research, Charlotte, North Carolina
  - Javara, Charlotte, North Carolina
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Clinical Trials of America, LLC, Mount Airy, North Carolina
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Great Lakes Medical Research, LLC, Beachwood, Ohio
  - Gastro Health Research, Cincinnati, Ohio
  - Hightop Medical Research Clinic, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dayton Clinical Resesarch, Dayton, Ohio
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Comprehensive Internal Medicine, Inc, Wooster, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - SSM Health Medical Group/Hightower Clinical, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Richard M. Kastelic, M.D., and Associates, P.C., Johnstown, Pennsylvania
  - Regional GI, Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Care Access Research, Pottsville, Pottsville, Pennsylvania
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - Invocare Medical Research & Healthcare Center, West Columbia, South Carolina
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Clinical Research Solutions, LLC - TN, Jackson, Tennessee
  - Tri-Cities, Kingsport, Tennessee
  - Great Lakes Medical Research, LLC, Union City, Tennessee
  - ARC Clinical Research at Four Points, Austin, Texas
  - Elligo Health Research Inc., Austin, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - Avant Research Associates, Austin, Texas
  - Mercy Family Clinic, Dallas, Texas
  - Dharma PA D/B/A Southwest Family Medicine Associates, Dallas, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Houston Digestive Disease, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Fairway Medical Clinic, Houston, Texas
  - Digestive System Healthcare, Houston, Texas
  - FMC Science, LLC, Lampasas, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Wellness Clinical Research, McKinney, Texas
  - ARC Clinical Research at Kelly Lane, Pflugerville, Texas
  - Epic Medical Research, LLC, Red Oak, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Progressive Clinical Research, LLC, Bountiful, Utah
  - Tanner Clinic, Layton, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Clinical Research, Riverton, Utah
  - Granger Medical Clinic, Riverton, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Summit Clinical Research, Petersburg, Virginia
  - Central Virginia VA Healthcare System, Richmond, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Spokane Gastroenterology, Spokane, Washington
  - Wenatchee Valley Hospital, Wenatchee, Washington
  - University Physicians and Surgeons, Inc. DBA Marshall Health, Huntington, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Ascension Wisconsin, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study may be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan, and informed consent form may also be shared. Data may be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data may be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research.

REFERENCES:
- [Derived] Imperiale TF, Gagrat ZD, Krockenberger M, Porter K, Ziegler E, Leduc CM, Matter MB, Olson MC, Limburg PJ. Algorithm Development and Early Performance Evaluation of a Next-Generation Multitarget Stool DNA Screening Test for Colorectal Cancer. Gastro Hep Adv. 2024 May 17;3(6):740-748. doi: 10.1016/j.gastha.2024.05.002. eCollection 2024. PMID 39280922
- [Derived] Imperiale TF, Porter K, Zella J, Gagrat ZD, Olson MC, Statz S, Garces J, Lavin PT, Aguilar H, Brinberg D, Berkelhammer C, Kisiel JB, Limburg PJ; BLUE-C Study Investigators. Next-Generation Multitarget Stool DNA Test for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):984-993. doi: 10.1056/NEJMoa2310336. PMID 38477986
- [Derived] Gagrat ZD, Krockenberger M, Bhattacharya A, Gagrat BZ, Leduc CM, Matter MB, Fourrier KD, Mahoney DW, Edwards V DK, Lidgard GP, Limburg PJ, Johnson SC, Domanico MJ, Kisiel JB. Next-generation Multi-target Stool DNA Panel Accurately Detects Colorectal Cancer and Advanced Precancerous Lesions. Cancer Prev Res (Phila). 2024 Mar 4;17(3):119-126. doi: 10.1158/1940-6207.CAPR-23-0285. PMID 38224564